CLINICAL TRIAL: NCT02287467
Title: Anti-Influenza Hyperimmune Intravenous Immunoglobulin Clinical Outcome Study (INSIGHT 006: FLU-IVIG)
Brief Title: Evaluating the Safety and Efficacy of Anti-Influenza Intravenous Hyperimmune Immunoglobulin (IVIG) in Adults Hospitalized With Influenza
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: University of Minnesota (Other); International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INSIGHT 006: FLU-IVIG
Record Dates: First submitted 2014-11-06; First posted 2014-11-10 (Estimated); Results first posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Influenza A; Influenza B
Keywords: Antiviral; IVIG; Hemagglutination inhibition (HAI); Antibody
MeSH Terms: interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: hIVIG (Experimental): Participants will receive a single infusion of intravenous hyperimmune immunoglobulin (hIVIG), administered over approximately 2 hours on Day 0. Participants will also receive SOC treatment for the flu.
  Interventions: Biological: Intravenous hyperimmune immunoglobulin (IVIG)
- Arm B: Placebo (Placebo Comparator): Participants will receive a single infusion of placebo for hIVIG, administered over approximately 2 hours on Day 0. Participants will also receive SOC treatment for the flu.
  Interventions: Biological: Placebo for IVIG

INTERVENTIONS:
Biological: Intravenous hyperimmune immunoglobulin (IVIG) — Administered intravenously (IV) at a dose of 0.25 g/kg (up to a maximum of 24.75 g, corresponding to approximately 100 kg actual body weight)
  Arms: Arm A: hIVIG
Biological: Placebo for IVIG — Administered IV as 500 mL of normal saline
  Arms: Arm B: Placebo

SUMMARY:
Influenza (the flu) is a common illness that usually occurs in autumn and winter. The flu is usually mild, but can cause serious illness or death. The purpose of this study is to test the safety and effectiveness of an antibody against the flu (called intravenous hyperimmune immunoglobulin or IVIG) in people who are hospitalized for severe flu.

DETAILED DESCRIPTION:
Influenza is responsible for thousands of hospitalizations and deaths each year in the United States and worldwide. One possible new treatment for the flu involves the use of IVIG, a blood product containing antibodies from people who have recovered from the flu or who have had a flu shot. The purpose of this study is to evaluate whether IVIG can reduce the severity and duration of flu in people who are hospitalized with the flu.

The study will enroll participants 18 years and older who are hospitalized with the flu. The study will enroll participants over one or more flu seasons. Regardless of the date of enrollment, each participant will be in the study for about 28 days.

At study entry (Day 0), participants will be randomly assigned to one of two groups (Arms A and B). Participants in both groups will receive standard of care (SOC) treatment for the flu, but those in Arm A will also receive one dose of IVIG and those in Arm B will receive a placebo for IVIG. Both IVIG and placebo will be given intravenously over at least 2 hours.

On Day 0, before receiving IVIG or placebo, participants will undergo a symptoms assessment, blood collection, and a nasopharyngeal (NP) swab to collect a sample of secretions from the nose and throat.

Additional study visits will occur on Days 1, 2, 3, 7, 14, and 28. Depending on the visit, participants may take part in the same study procedures that took place on Day 0. On Days 2, 14, and 28, visits for participants who are no longer hospitalized may be conducted over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Locally determined positive influenza test (by polymerase chain reaction [PCR] or other nucleic acid test, or by rapid antigen [Ag]) from a specimen obtained within 2 days prior to randomization
* Onset of illness no more than 7 days before randomization, defined as when the participant first experienced at least one respiratory symptom or fever
* Hospitalized (or in observation unit) for influenza, with anticipated hospitalization for more than 24 hours. Criteria for hospitalization will be up to the individual treating clinician.
* For women of child-bearing potential: willingness to abstain from sexual intercourse or use at least one form of hormonal or barrier contraception through Day 28 of the study
* Willingness to have blood and respiratory samples obtained and stored
* NEW score greater than or equal to 2 at screening (see the protocol for more information on this criterion)

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Strong clinical evidence (in the judgment of the site investigator) that the etiology of illness is primarily bacterial in origin
* Prior treatment with any investigational drug therapy within 30 days prior to screening
* History of allergic reaction to blood or plasma products (as judged by the site investigator)
* Known immunoglobulin A (IgA) deficiency
* A pre-existing condition or use of a medication that, in the opinion of the site investigator, may place the participant at a substantially increased risk of thrombosis (e.g., cryoglobulinemia, severe refractory hypertriglyceridemia, or clinically significant monoclonal gammopathy)
* Presence of any pre-existing illness that, in the opinion of the site investigator, would place the participant at an unreasonably increased risk through participation in this study
* Participants who, in the judgment of the site investigator, will be unlikely to comply with the requirements of this protocol
* Medical conditions for which receipt of a 500 mL volume of intravenous fluid may be dangerous to the participant (e.g., decompensated congestive heart failure)
* Receiving extracorporeal membrane oxygenation (ECMO)
* Suspicion that infection is due to an influenza strain or subtype other than A(H1N1)pdm09, H3N2, or influenza B (e.g., H5N1, H7N9)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2015-01; Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T. Davey, Jr., MD, Study Chair — National Institute of Allergy and Infectious Diseases (NIAID); Eduardo Fernández-Cruz, MD, PhD, Study Chair — Hospital General Universitario Gregorio Marañón; Norman P. Markowitz, MD, Study Chair — The Henry Ford Hospital; Sarah L. Pett, MD, MBBS, DTM, MRCP (UK), Study Chair — University College, London
Locations (21):
- United States (17):
  - UCSD Antiviral Research Center (A VRC), San Diego, California
  - Denver Public Health, Denver, Colorado
  - University of Illinois, Chicago, Illinois
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Cooper University Hospital, Camden, New Jersey
  - Cornell CRS, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - OHIO State University (OSU) Wexner Medical Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - West Virginia University, Morgantown, West Virginia
- Westmead Hospital, Sydney, Australia
- Odense University Hospital, Odense, Denmark
- United Kingdom (2):
  - St James's University Hospital, Leeds
  - Churchill Hospital, Oxford

REFERENCES:
- [Derived] Vanderven HA, Wentworth DN, Han WM, Peck H, Barr IG, Davey RT Jr, Beigel JH, Dwyer DE, Jain MK, Angus B, Brandt CT, Mykietiuk A, Law MG, Neaton JD, Kent SJ; INSIGHT FLU-IVIG Study Group. Understanding the treatment benefit of hyperimmune anti-influenza intravenous immunoglobulin (Flu-IVIG) for severe human influenza. JCI Insight. 2023 Jul 24;8(14):e167464. doi: 10.1172/jci.insight.167464. PMID 37289541
- [Derived] Davey RT Jr, Fernandez-Cruz E, Markowitz N, Pett S, Babiker AG, Wentworth D, Khurana S, Engen N, Gordin F, Jain MK, Kan V, Polizzotto MN, Riska P, Ruxrungtham K, Temesgen Z, Lundgren J, Beigel JH, Lane HC, Neaton JD; INSIGHT FLU-IVIG Study Group. Anti-influenza hyperimmune intravenous immunoglobulin for adults with influenza A or B infection (FLU-IVIG): a double-blind, randomised, placebo-controlled trial. Lancet Respir Med. 2019 Nov;7(11):951-963. doi: 10.1016/S2213-2600(19)30253-X. Epub 2019 Sep 30. PMID 31582358

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: hIVIG: Participants will receive a single infusion of intravenous hyperimmune immunoglobulin (IVIG), administered over approximately 2 hours on Day 0. Participants will also receive standard of care (SOC )treatment for the flu.
  Intravenous hyperimmune immunoglobulin (IVIG): Administered intravenously (IV) at a dose of 0.25 g/kg (up to a maximum of 24.75 g, corresponding to approximately 100 kg actual body weight)
- Arm B: Placebo: Participants will receive a single infusion of placebo for IVIG (saline), administered over approximately 2 hours on Day 0. Participants will also receive SOC treatment for the flu.
  Placebo for IVIG: Administered IV as 500 mL of normal saline
Period: Overall Study
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Started | 168 | 161
Completed | 156 | 152
Not Completed | 12 | 9
Not completed — Protocol Violation | 12 | 9

BASELINE CHARACTERISTICS:
Population: Participants in the analysis data set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: hIVIG | Arm B: Placebo | Total
Number analyzed (Participants) | 156 | 152 | 308
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 109 | 100 | 209
  >=65 years | 46 | 51 | 97
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [41 to 68] | 57 [48 to 68] | 57 [45 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 88 | 168
  Male | 76 | 64 | 140
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Asian | 33 | 36 | 69
  Race/ethnicity: Black/African American | 27 | 30 | 57
  Race/ethnicity: Hispanic | 27 | 24 | 51
  Race/ethnicity: White/Caucasian | 67 | 61 | 128
  Race/ethnicity: Other | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 91 | 84 | 175
  United Kingdom | 8 | 10 | 18
  Australia | 5 | 5 | 10
  Argentina | 4 | 4 | 8
  Denmark | 5 | 3 | 8
  Spain | 5 | 5 | 10
  Greece | 5 | 4 | 9
  Mexico | 1 | 2 | 3
  Thailand | 32 | 35 | 67
National Early Warning (NEW) score [Median (Inter-Quartile Range); unit: units on a scale] — National Early Warning score measured on day of randomization. The NEW score is a morbidity index based on 6 vital signs (respiratory rate, oxygen saturation, temperature, blood pressure, pulse/heart rate, level of consciousness). Each component is scored from 0 to 3 (best to worst) and the components are summed. Thus the composite score can range from 0 to 18.
  units on a scale | 4 [2 to 6] | 4 [2 to 6] | 4 [2 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Each of 6 Clinical Status Categories on Day 7
Description: This is the primary outcome, a 6-category ordinal outcome ranging from death (worst) to discharged from hospital with resumption of normal activities (best).
Time Frame: Assessed on Day 7
Population: All infused participants, using multiple imputation to impute outcome for 4 participants with missing data.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: hIVIG: Participants will receive a single infusion of intravenous hyperimmune immunoglobulin (IVIG), administered over approximately 2 hours on Day 0. Participants will also receive SOC treatment for the flu.
  Intravenous hyperimmune immunoglobulin (IVIG): Administered intravenously (IV) at a dose of 0.25 g/kg (up to a maximum of 24.75 g, corresponding to approximately 100 kg actual body weight)
- Arm B: Placebo: Participants will receive a single infusion of placebo for IVIG, administered over approximately 2 hours on Day 0. Participants will also receive SOC treatment for the flu.
  Placebo for IVIG: Administered IV as 500 mL of normal saline
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 156 | 152
Participants
  Died | 3 | 2
  Hospitalized, in ICU | 6 | 11
  Non-ICU hospitalization, using supplemental oxygen | 15 | 16
  Non-ICU hospitalization, no supplemental oxygen | 8 | 12
  Discharged, not back to normal activities | 56 | 51
  Discharged, back to normal activities | 68 | 60
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Odds ratio of being in a better category, as assessed using a proportional odds model. Multiple imputation techniques were used to impute an outcome for 4 patients for whom the outcome was unknown; Test type: Superiority; p = .33, Regression, Logistic; Adjusted for baseline clinical status, region, and participation in the pilot study; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.79 to 1.97] — Odds ratio is hIVIG vs. placebo. A value greater than 1 favors the hIVIG group

2. Secondary Outcome: Number of Patients in Each of 5 Clinical Status Categories on Day 3
Description: 5-category ordinal outcome assessed on day 3; clinical status ranges from death (worst) to discharged from the hospital (best).
Time Frame: Assessed on Day 3
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 156 | 152
Participants
  Death | 1 | 0
  Hospitalized, in ICU | 8 | 13
  Non-ICU hospitalization, NEW score 3+ | 25 | 31
  Non-ICU hospitalization, NEW score < 3 | 55 | 46
  Discharged | 67 | 62
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Odds ratio for being in a better category, from a proportional odds model; Test type: Superiority; p = .84, Regression, Logistic; Adjusted for baseline clinical status, region, and participation in the pilot study; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.61 to 1.48] — Odds ratio is for hIVIG vs placebo. An odds ratio greater than 1 favors the hIVIG group

3. Secondary Outcome: Number of Patients in Each of 6 Clinical Status Categories on Day 3
Description: 6-category ordinal outcome evaluated on Day 3; clinical status ranges from death (worst) to discharged from hospital with resumption of normal activities (best).
Time Frame: Measured on Day 3
Population: All participants with clinical data available on Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 155 | 152
Participants
  Death | 1 | 0
  Hospitalized, in ICU | 8 | 13
  Non-ICU hospitalization, on supplemental oxygen | 37 | 34
  Non-ICU hospitalizaiton, no supplemental oxygen | 43 | 43
  Discharged, not back to normal activities | 53 | 53
  Discharged, back to normal activities | 13 | 9
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Odds ratio for being in a better group, from a proportional odds model; Test type: Superiority; p = .52, Regression, Cox; adjusted for baseline clinical status, region, and participation in the pilot study; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.57 to 1.33] — Odds ratio is for hIVIG vs. placebo. An odds ratio > 1 favors the hIVIG group

4. Secondary Outcome: Number of Patients With a Favorable Outcome on Day 7
Description: Sliding dichotomy defined as non-ICU hospitalization or discharge if enrolled from ICU, and discharge if enrolled from the general ward.
Time Frame: Assessed on Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 156 | 152
Participants
  favorable outcome | 128 | 115
  unfavorable outcome | 28 | 37
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Test type: Superiority; p = .20, Regression, Logistic; adjusted for baseline clinical status, region, and participation in the pilot study; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.81 to 2.74] — Odds ratio for hIVIG vs placebo. An odds ratio > 1.0 favors the hIVIG group

5. Secondary Outcome: Hospital Discharge
Description: Number of participants alive and discharged from the hospital
Time Frame: Measured through Day 7
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 156 | 152
Participants
  Discharged alive | 119 | 110
  Not discharged alive | 37 | 42
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Deaths during hospitalization are censored after day 7; Test type: Superiority; p = .44, Regression, Cox; Stratified by baseline clinical status, region, and participation in the pilot study; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [.85 to 1.45] — hazard ratio is hIVIG vs placebo; a hazard ratio >1 favors the hIVIG group

6. Secondary Outcome: Mortality
Description: Number of participants dying through day 28.
Time Frame: Measured through day 28
Population: all participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 156 | 152
Participants
  Died | 6 | 5
  Did not die | 150 | 147
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Test type: Superiority; p = .40, Regression, Cox; stratified by baseline clinical status, region, and participation in pilot study; Hazard Ratio (HR) = 1.72, 95% CI 2-sided [.48 to 6.15] — hazard ratio is for hIVIG vs placebo; a hazard ratio < 1.0 favors the hIVIG group

7. Secondary Outcome: Number of Patients Alive and Out of Hospital
Description: Number and percent alive and out of hospital on day 28
Time Frame: Measured through Day 28
Population: All participants with vital status known on Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 155 | 151
Participants
  Alive and out of hospital | 140 | 137
  Died or hospitalized | 15 | 14
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Test type: Superiority; p = .74, Regression, Logistic; adjusted for baseline clinical status, region, and participation in pilot study; Odds Ratio (OR) = 0.87, 95% CI 2-sided [.38 to 1.98] — odds ratio is for hIVIG vs placebo; an odds ratio > 1.0 favors hIVIG

8. Secondary Outcome: Change in Viral Load
Description: Change in nasopharyngeal viral load from baseline to day 3
Time Frame: Day 3
Population: Participants with viral load results at both baseline and day 3. Participants with undetectable viral load results at baseline are excluded.
Measure: Mean (Standard Error); unit: log10 RNA
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 134 | 136
log10 RNA | -1.99 (.16) | -2.32 (.17)
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Test type: Superiority; p = .49, Regression, Linear; Adjusted for baseline RNA, geographic region, and influenza subtype; Mean Difference (Net) = 0.14, 95% CI 2-sided [-.26 to .54] — Change is calculated as day 3 - baseline. Difference in changes is hIVIG - placebo

9. Secondary Outcome: Death or Re-hospitalization
Description: Number and percent of participants who died or were re-hospitalized after initial discharge
Time Frame: Day 28
Population: all participants with data
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 150 | 146
Participants | 19 | 19
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Test type: Superiority; p = .93, Regression, Logistic; adjusted for baseline clinical status, region, and participation in pilot study; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.5 to 1.97] — Odds ratio is for hIVIG vs placebo

10. Secondary Outcome: Percent of Participants Developing Complications
Description: Number and percent of participants developing respiratory distress syndrome, acute renal failure, sepsis, pneumonia, enteritis, or bronchitis
Time Frame: Measured through Day 28
Population: all participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 156 | 152
Participants | 20 | 22
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Test type: Superiority; p = .81, Regression, Logistic; adjusted for baseline clinical status, region, and participation in pilot study; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.5 to 1.82] — odds ratio is for hIVIG group vs placebo

11. Secondary Outcome: Number of Patients in Each of 6 Clinical Status Categories on Day 14
Description: 6-category ordinal outcome measured on day 14
Time Frame: Measured on day 14
Population: participants with observed data on day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 152 | 151
Participants
  Died | 4 | 4
  Hospitalized in ICU | 5 | 6
  Hospitalized on supplement oxygen | 8 | 5
  Hospitalized not on supplemental oxygen | 4 | 11
  Discharged, not back to normal activities | 29 | 33
  Discharged, back to normal activities | 102 | 92
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Proportional odds for being in a better category; Test type: Superiority; p = .55, Regression, Logistic; adjusted for baseline clinical status, region, and participation in the pilot study; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.70 to 1.95] — Odds ratio (hIVIG vs placebo) of being in a better category. An odds ratio > 1 favors the hIVIG group

12. Secondary Outcome: Number of Patients Alive and Out of Hospital on Day 14
Description: Number and percentage of participants alive and out of the hospital on Day 14
Time Frame: day 14
Population: all participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 155 | 151
Participants | 134 | 125
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Test type: Superiority; p = .77, Regression, Logistic; adjusted for baseline clinical status, region, and participation in pilot study; Odds Ratio (OR) = 1.12, 95% CI 2-sided [.5 to 2.31] — odds ratio is for hIVIG vs placebo

13. Secondary Outcome: Resumption of Normal Activities by Day 14
Description: Participants reporting resumption of normal daily activities by Day 14
Time Frame: day 14
Population: Participants with observed data
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 152 | 151
Participants | 102 | 92
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Test type: Superiority; p = .34, Regression, Logistic; adjusted for baseline clinical status, region, and participation in pilot study; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.7 to 2.34] — odds ratio is expressed as hIVIG vs placebo

14. Secondary Outcome: Number of Patients in Each of 6 Clinical Status Categories on Day 28
Description: 6-category ordinal outcome corresponding to clinical status on day 28
Time Frame: day 28
Population: participants with observed data
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 151 | 150
Participants
  Died | 6 | 5
  Hospitalized in ICU | 2 | 2
  Hospitalized, on supplemental oxygen | 6 | 2
  Hospitalized, not on supplemental oxygen | 1 | 5
  Discharged, not back to normal activities | 21 | 22
  Discharged, back to normal activities | 115 | 114
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Test type: Superiority; p = .73, Regression, Logistic — adjusted for baseline clinical status, region, and participation in pilot study; adjusted for baseline clinical status, region, and participation in pilot study; Odds Ratio (OR) = .90, 95% CI 2-sided [.50 to 1.62] — odds ratio (hIVIG vs placebo) is for being in a better category. An odds ratio >1 favors the hIVIG group

15. Secondary Outcome: Number of Influenza A-Infected Patients in Each of 6 Clinical Status Categories on Day 7
Description: Primary 6-category ordinal outcome for participants infected with Influenza A
Time Frame: Day 7
Population: all participants infected with influenza A
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 114 | 110
Participants
  Died | 3 | 0
  Hospitalized in ICU | 5 | 7
  Hospitalized on supplemental oxygen | 14 | 9
  Hospitalized not on supplemental oxygen | 7 | 10
  Discharged, not back to normal activities | 40 | 39
  Discharged, back to normal activities | 45 | 45
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Multiple imputation was used to estimate the outcome for 3 participants for whom the outcome was partially unknown; Test type: Superiority; p = .82, Regression, Logistic; adjusted for baseline clinical status, region, and participation in the pilot study; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.55 to 1.59] — Odds ratio (hIVIG vs placebo) is for being in a better category

16. Secondary Outcome: Number of Influenza B-Infected Patients in Each of 6 Clinical Status Categories on Day 7
Description: Primary 6-category ordinal outcome for subgroup of participants infected with influenza B
Time Frame: Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 42 | 42
Participants
  Died | 0 | 2
  Hospitalized in ICU | 1 | 4
  Hospitalized on supplemental oxygen | 1 | 7
  Hospitalized not on supplemental oxygen | 1 | 2
  Discharged, not back to normal activities | 16 | 12
  Discharged, back to normal activities | 23 | 15
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Multiple imputation was used to estimate the outcome for one participant; Test type: Superiority; p = .02, Regression, Logistic; adjusted for baseline clinical status, region, and participation in pilot study; Odds Ratio (OR) = 3.19, 95% CI 2-sided [1.21 to 8.42] — Odds ratio (hIVIG vs placebo) for a better outcome. An odds ratio > 1 favors the hIVIG group

17. Secondary Outcome: pH1N1 Titers at Day 7
Description: pH1N1 hemagglutination inhibition assay (HAI) titers among participants infected with pH1N1 using A/Cal/2009 as reference virus
Time Frame: Day 7
Population: participants infected with pH1N1 with HAI titers measured at day 7
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 23 | 26
titer | 285 (374) | 229 (341)
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; HAI measurements were log-transformed to compute treatment differences and the model was adjusted for baseline titer; Test type: Superiority; p = .18, Mixed Models Analysis; longitudinal regression with adjustment for baseline titer; ratio of geometric means = 1.50, 95% CI 2-sided [0.84 to 2.7] — Ratio of hIVIG group to placebo group. A ratio > 1.0 indicates higher titers for the hIVIG group

18. Secondary Outcome: H3N2 Titers at Day 7
Description: H3N2 HAI titers among participants infected with H3N2 using A/HongKong/2014 as reference virus
Time Frame: Day 7
Population: participants infected with H3N2 with HAI titers measured at day 7
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 54 | 49
titer | 259 (291) | 225 (277)
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Test type: Superiority; p = .13, Mixed Models Analysis; longitudinal analysis of log-transformed titers adjust for baseline titer; ratio of geometric means = 1.31, 95% CI 2-sided [0.93 to 1.8] — Ratio of geometric means of hIVIG vs placebo. A ratio >1.0 indicates higher titers in the hIVIG group on day 7

19. Secondary Outcome: Influenza B Titers at Day 7
Description: Flu B HAI titers among participants infected with influenza B using B/Phuket/2013 as reference virus
Time Frame: Day 7
Population: participants infected with influenza B with HAI titers measured at day 7
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | Arm A: hIVIG | Arm B: Placebo
Number analyzed (Participants) | 39 | 40
titer | 112 (161) | 84 (83)
Statistical Analysis 1: Comparison: Arm A: hIVIG vs Arm B: Placebo; Test type: Superiority; p = .78, Mixed Models Analysis; log-transformed titers adjusted for baseline titer; ratio of geometric means = 0.94, 95% CI 2-sided [0.58 to 1.5] — ratio of geometric mean for hIVIG vs placebo. A ratio > 1.0 indicates higher titers at day 7 for the hIVIG group

ADVERSE EVENTS:
Time Frame: 28 days
Description: Serious adverse events plus all grade 3 and 4 adverse events, as graded according to the National Institute of Health Division of AIDS (DAIDS) toxicity table.
Arm/Group | Arm A: hIVIG | Arm B: Placebo
All-Cause Mortality (participants affected / at risk) | 6/156 | 5/152
Serious Adverse Events (participants affected / at risk) | 25/156 | 26/152
Other Adverse Events (participants affected / at risk) | 13/156 | 14/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: hIVIG (N=156) | Arm B: Placebo (N=152)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Internal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 1 (1)
Dysthymic disorders (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: hIVIG (N=156) | Arm B: Placebo (N=152)
Blood creatinine increased (Investigations) | 4 (5) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Haemoglobin decreased (Investigations) | 2 (4) | 4 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT02287467/SAP_000.pdf
  • Study Protocol (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT02287467/Prot_001.pdf